CLINICAL TRIAL: NCT00792740
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of ITF2357 on Mucosal Healing in Patients With Moderate-to-severe Active Crohn's Disease
Brief Title: Effect of ITF2357 on Mucosal Healing in Patients With Moderate-to-severe Active Crohn's Disease
Acronym: CD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: As no safety warnings were detected, Interim analysis from the first 40 patients recommends to stop the trial for futility
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSC/06/2357/23; 2007-000189-19 (EudraCT Number)
Record Dates: First submitted 2008-11-14; First posted 2008-11-18 (Estimated); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2022-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — givinostat hydrochloride; givinostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Oral matching placebo capsules, administered bid.
  Interventions: Other: Placebo
- ITF2357 (Experimental): Oral ITF2357 50 mg bid
  Interventions: Drug: ITF2357

INTERVENTIONS:
Drug: ITF2357 — ITF2357 was administered as hard gelatin capsules for oral administration at the dose strength of 50 mg. Capsules were administered as follow: one capsule in the morning and one in the evening.
  Other Names: Givinostat
  Arms: ITF2357
Other: Placebo — Placebo was supplied as matching capsules for oral administration with the same outer appearance of the study drug and with the same dosing scheme (one capsule in the morning and one in the evening)
  Arms: Placebo

SUMMARY:
Objectives:

The primary objective of the study was to determine the ability of ITF2357, administered orally at the dose of 50 mg b.i.d. for 8 consecutive weeks, to induce complete healing of mucosal ulcerations of ileum and/or colon, assessed by endoscopy, in patients with endoscopic and clinical evidence of active moderate-to-severe Crohn's disease not controlled by conventional therapies.

The secondary objectives of the study were:

* to evaluate the effect of ITF2357 on endoscopic disease activity assessed using both the Crohn's Disease Endoscopic Index of Severity (CDEIS) and the Simple Endoscopic Score of Crohn's Disease (SES-CD);
* to evaluate the effect of ITF2357 on clinical disease activity, assessed using the Crohn's Disease Activity Index (CDAI);
* to assess the safety and tolerability of ITF2357; to assess the pharmacokinetic profile of ITF2357.

DETAILED DESCRIPTION:
The study was conducted according to a randomized, double-blind placebo-controlled, parallel group design in up to 25 clinical sites in Europe.

Eligible patients were randomly assigned to two parallel treatment groups (1:1 randomization ratio) receiving either ITF2357, as hard gelatine capsule for oral administration, at the dose of 50 mg b.i.d. (total daily dose of 100 mg), or matching placebo capsules.

Treatment was administered on an outpatient basis for 8 consecutive weeks, followed by a 4-week follow-up.

During screening, in the 8-week treatment period and in the 4-week follow-up period, patients attended scheduled visits, with physical and laboratory assessments, in order to monitor disease evolution and safety and tolerability of ITF2357.

The study was planned to be conducted in up to 80 patients of both genders, with established diagnosis of CD, who presented with ulcerations greater than aphthous ulcers in at least one of the five bowel segments investigated endoscopically, from the ileum to the rectum, with endoscopic and clinical evidence of moderate-to-severe active disease, not controlled by on-going treatment with conventional therapies such as 5-aminosalicylates, steroids or immunosuppressants.

The present study has been designed in order to assessed wether short-term (8 weeks) treatment with oral ITF2357 can induce disease improvement in a substantial proportion of patients.

Its aim to evaluate whether a short term treatment with ITF2357 for 8 weeks, at the selected dose of 50 mg b.i.d., is able to induce healing of mucosal lesions, evaluated endoscopically, in patients with endoscopic and clinical evidence of moderate-to-severe active Crohn's disease, not controlled by ongoing treatment with conventional therapies such as 5-aminosalicylates, steroids or immunosuppressants, was not addressed and the study was prematurely interrupted according to IDSMC (Independent Data and Safety Monitoring Committee) decision, based on the results of the interim analysis, which did not demonstrate any benefit of ITF2357 over placebo in the primary variable rate of patients achieving complete healing at week 8.

There was also no evidence of benefits in patients treated with ITF2357 compared to placebo in the secondary efficacy endpoints (full remission rate, remission rate, CDEIS endoscopic response, changes from baseline of CDEIS score and SES-CD score, changes from baseline of CDAI score, CDAI remission rate, and CDAI response rate).

ELIGIBILITY:
Inclusion Criteria:

* Age: > 18 years
* Diagnosis of CD, re-established by endoscopy and/or X-ray and/or surgery in the last 36 months
* CD in active phase since at least 2 weeks before screening
* CDAI between 220 and 450
* CDEIS > 8
* Ulcerations greater than aphthous ulcers in at least 1 of the bowel segments from ileum to rectum
* If any on-going treatment with corticosteroids (prednisone, prednisolone or budesonide), it must be at a dose equivalent to or less than 30 mg/day prednisone, or 9 mg of budesonide, and in use for at least one month and at a stable dose for at least two weeks before patient enrolment
* If any on-going treatment with immunosuppressant (azathioprine, 6-mercaptopurine, methotrexate), it must be in use for at least 3 months before patient enrolment
* If any on-going treatment with 5-aminosalicylates, it must be in place for at least 4 weeks before patient enrolment, at a dose > 2 g
* Females of childbearing potential with negative pregnancy tests
* Signed written informed consent to participate in this trial.

Exclusion Criteria:

* Treatment in the 2 months with anti-TNF-alfa antibodies and in the previous 3 months with cytokines inhibitors or experimental drugs
* Primary failure to previous treatment with anti-TNF-alfa antibodies-
* Current bowel obstruction or any condition that may predispose to its development (e.g. clinically significant unresolved intestinal stricture, adhesions or any other condition that would place the patient at risk for developing overt bowel obstruction) or intestinal perforation or significant GI hemorrhage
* Expected surgery for the duration of the study
* Any ostomy or extensive bowel resection
* Positive serological anti-HCV and anti-HIV testing and positive testing for active HBV replication, e.g. HBV-DNA or HBsAg or HBeAg (to be performed at screening)
* Other on-going clinical relevant viral infections (e.g. herpes zoster, Epstein-Barr, CMV), systemic fungal infections or history of recurrent serious bacterial infections
* Signs and symptoms of severe, progressive or uncontrolled renal, hepatic, haematologic, endocrine, pulmonary, cardiac, neurologic or cerebral disease
* Any previous evidence, irrespective of its severity, of coronary disease, cardiac rhythm abnormalities or congestive heart failure
* QTc interval > 450 msec at pre-treatment evaluation
* Serum magnesium and potassium below the LLN at pre-treatment evaluation
* Platelet counts below 200 x 10^9/L at pre-treatment evaluation
* Any previous evidence, irrespective of its severity, of renal function impairment
* Unavoidable concomitant treatment with any drug known for potential risk of causing Torsades de Pointes
* Presence of a transplanted organ
* History of cancer with less than 5 years documentation of a disease-free state
* History of tuberculosis
* Severe lactose intolerance
* Pregnant or nursing women
* Female of childbearing potential without using a safe contraceptive measure
* Participation in a clinical trial within 30 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-10-22 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2009-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Rutgeerts, MD, Study Chair — University Hospital Gasthuisberg, Leuven, Belgium
Locations (10):
- Belgium (6):
  - AZ Sint Lucas Gastro-enterologie, Assebroek
  - Imelda Hospital Gastro-enterology dept., Bonheiden
  - CHU Saint-Pierre Médecine Interne, Brussels
  - UZ Gent Gastro-enterologie 1K12IE, Ghent
  - AZ Groeninge (St-Niklaas) Gastro-enterologie, Kortrijk
  - University Hospital Gasthuisber, Leuven
- Divisione di Gatroenterologia Istituto Clinico Humanitas IRCCS in. Gastroenterology, Rozzano, Italy
- Netherlands (3):
  - Vrije Universiteit (VU) Medisch Centrum Afdeling M.D.L.ziekten, Amsterdam
  - Academisch Medisch Centrum (AMC) Afdeling M.D.L. ziekten, Amsterdam
  - Leids Universitair Medisch Centrum (LUMC) Afdeling M.D.L. ziekten, Leiden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty-one (51) subjects were enrolled in the study, as planned, and 37 of them completed the study as per protocol.
Groups:
- Placebo: Oral matching placebo capsules, administered bid.
  Placebo: Placebo will be supplied as matching capsules for oral administration with the same outer appearance of the study drug and with the same dosing scheme (one capsule in the morning and one in the evening)
Period: Overall Study
Arm/Group | Placebo | ITF2357
Started | 26 | 25
Completed | 19 | 18
Not Completed | 7 | 7
Not completed — Disease Worsening | 3 | 2
Not completed — Personal Reason | 1 | 0
Not completed — Adverse Event | 1 | 3
Not completed — Patient's withdrawal of consent | 0 | 1
Not completed — Termination of the trial by the Sponsor | 2 | 0
Not completed — Other reasons | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT: All randomized patients who received at least one treatment with study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ITF2357 | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 24 | 50
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 25 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Complete Healing of Mucosal Ulcerations of Ileum and/or Colon
Description: The outcome is assessed by endoscopy, in patients with endoscopic and clinical evidence of active moderate-to-severe Crohn's disease not controlled by conventional therapies.
  The outcome measure defines the rate of patients achieving complete healing in ITT population, i.e disappearance of mucosal ulceration, obtained with ITF2357 treatment.
Time Frame: At week 8
Population: ITT: population included all randomized patients who took at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ITF2357
Number analyzed (Participants) | 26 | 25
Participants | 0 | 1

2. Secondary Outcome: Number of Patients Achieving Full Endoscopic Remission ( Based on CDEIS Score)
Description: CDEIS (Crohn's Disease Endoscopic Index of Severity) is an index for determining the severity of Crohn's disease with endoscopic localization to ileum and colon; A patient was defined 'fully endoscopic remissed' whether the CDEIS score at week 8 was equal or lower than three points
  CDEIS score considers 4 parameters, each one evaluated in 5 pre-defined segments of the colon.
  The score can be calculated even in case of incomplete investigations, as the results of the individual segments are divided by the number of segments investigated.
  Score Scale:
  < 3 remission; 3 - 8 mild endoscopic activity; 9 - 12 moderate endoscopic activity; > 12 severe endoscopic activity.
  The higher the score, the worse is patient's situation.
Time Frame: At Week 8
Population: ITT population included all randomized patients who took at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ITF2357
Number analyzed (Participants) | 26 | 25
Participants | 2 | 1

3. Secondary Outcome: Number of Patients Achieving Endoscopic Remission (Based on CDEIS Score)
Description: CDEIS (Crohn's Disease Endoscopic Index of Severity) is an index for determining the severity of Crohn's disease with endoscopic localization to ileum and colon; A patient was defined 'endoscopic remissed' whether the CDEIS score at week 8 was equal or lower than six points.
  CDEIS score considers 4 parameters, each one evaluated in 5 pre-defined segments of the colon ).
  The score can be calculated even in case of incomplete investigations, as the results of the individual segments are divided by the number of segments investigated.
  The higher the score, the worse is patient's situation.
  Score Scale:
  < 3 remission; 3 - 8 mild endoscopic activity; 9 - 12 moderate endoscopic activity; > 12 severe endoscopic activity.
  A patient was defined 'endoscopic remissed' whether the CDEIS score at week 8 was equal or lower than six points.
Time Frame: At week 8
Population: ITT population included all randomized patients who took at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ITF2357
Number analyzed (Participants) | 26 | 25
Participants | 3 | 5

4. Secondary Outcome: Number of Patients Achieving Endoscopic Response (Based on CDEIS Score)
Description: CDEIS (Crohn's Disease Endoscopic Index of Severity) is an index for determining the severity of Crohn's disease with endoscopic localization to ileum and colon;
  A patient was considered in 'endoscopic response' whether the change in CDEIS score at week 8 versus baseline was equal or greater than 4.5 points.
  CDEIS score considers 4 parameters, each one evaluated in 5 pre-defined segments of the colon ).
  The score can be calculated even in case of incomplete investigations, as the results of the individual segments are divided by the number of segments investigated.
  The higher the score, the worse is patient's situation
  Score Scale:
  < 3 remission; 3 - 8 mild endoscopic activity; 9 - 12 moderate endoscopic activity; > 12 severe endoscopic activity.
  A patient was considered in 'endoscopic response' whether the change in CDEIS score at week 8 versus baseline was equal or greater than 4.5 points.
Time Frame: At week 8
Population: ITT population included all randomized patients who took at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ITF2357
Number analyzed (Participants) | 26 | 25
Participants | 6 | 7

5. Secondary Outcome: The Mean Changes of Crohn's Disease Endoscopic Index of Severity (CDEIS) From Baseline to Week 8
Description: CDEIS is an index to determ the endoscopic severity of Crohn's disease. Its score considers 4 parameters, each one evaluated in 5 pre-defined segments of the colon (ileum, ascending colon, transverse colon, descending colon and sigmoid loop, and rectum). These 4 parameters are: Deep ulcerations (12 if present, 0 if absent = total 1); Superficial ulcerations (6 if present, 0 if absent = total 2); Surface involved by disease (mm/10 on VAS = = total 3); Surface involved by ulcerations (mm/10 on VAS = total 4).
  Sum of Totals 1+2+3+4 =Total A Number of segments visualized in part or entirely (from 1 to 5)= n Total A/n =Total B if ulcerated stenosis in any segment, add 3 =Total C If non-ulcerated stenosis in any segment, add 3= Total D Total B+C+D=CDEIS grand score (min=0; max=NA)
  Decoding score < 3 remission; 3 - 8 mild endoscopic activity; 9 - 12 moderate endoscopic activity; > 12 severe endoscopic activity.
  The higher the score, the worse is patient's status.
Time Frame: From Baseline to week 8
Population: ITT population included all randomized patients who took at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | ITF2357
Number analyzed (Participants) | 26 | 25
score on a scale | -2.5 (5.6) | -2.4 (4.2)

6. Secondary Outcome: The Mean Changes of Simple Endoscopic Score for Crohn Disease (SES-CD) From Baseline to Week 8
Description: SES-CD is another index to determ the endoscopic severity of Crohn's disease. Its score considers 4 parameters, each one evaluated in 5 pre-defined segments of the colon (ileum, ascending colon, transverse colon, descending colon and sigmoid loop, and rectum). These 4 parameters are:
  ulcers? 0: no; 1: aphthous (0.1-0.5 cm); 2: large (0.5-2 cm); 3: very large (>2 cm); Surface involved by inflammation 0: 0%
  1: <50% 2: 50-75% 3: >75% Surface involved by ulcerations 0: 0%
  1. <10%
  2. 10-30%
  3. >30% Stenosis?
  0: No
  1. Single, can be passed
  2. Multiple, can be passed
  3. Cannot be passed The scores for each individual segment are added together as a sum score (min=0; max=60) The higher the score, the worse the outcome.
  Decoding score 0 - 2 remission 3 - 6 mild endoscopic activity 7 - 15 moderate endoscopic activity > 15 severe endoscopic activity
Time Frame: From Baseline to week 8
Population: ITT population included all randomized patients who took at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | ITF2357
Number analyzed (Participants) | 26 | 25
score on a scale | -2.6 (4.5) | -2.0 (4.0)

7. Secondary Outcome: The Mean Changes of CDAI Score From Baseline to Week 4-8-follow up
Description: CDAI (Crohn's Disease Activity Index): frequently used to assess disease severity. It gives a score ranging from 0 to over 600, based on a diary of symptoms kept by the patient for 7 days, and other measurements such as the patient's weight and haematocrit.
  The higher the score, the worse is patient's situation A patient is defined 'remissed' whether the CDAI score is lower than 150 points.
  A patient is defined 'responder' whether the change in CDAI score versus baseline is greater to 100 points
Time Frame: Weeks 4 and 8, and follow-up at 1 month
Population: ITT population included all randomized patients who took at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | ITF2357
Number analyzed (Participants) | 26 | 25
score on a scale
  At week 4 | -85.3 (95.9) | -32.7 (84.5)
  At week 8 | -119 (96.5) | -54.7 (94.3)
  At follow-up 1 month | -106 (91.6) | -83.8 (82.0)

8. Secondary Outcome: Number of Patients Achieving Remission (Based on CDAI Score)
Description: "Remission" is defined as the disappearance of signs and symptoms of the disease.
  CDAI (Crohn's Disease Activity Index): frequently used to assess disease severity. It gives a score ranging from 0 to over 600, based on a diary of symptoms kept by the patient for 7 days, and other measurements such as the patient's weight and haematocrit.
  The higher the score, the worse is patient's situation A patient is defined 'remissed' whether the CDAI score is lower than 150 points.
  A patient is defined 'responder' whether the change in CDAI score versus baseline is greater to 100 points
Time Frame: Weeks 4 and 8, and follow-up at 1 month
Population: ITT population included all randomized patients who took at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ITF2357
Number analyzed (Participants) | 26 | 25
Participants
  At week 4 | 10 | 4
  At week 8 | 14 | 7
  At follow-up after one month | 11 | 9

9. Secondary Outcome: Number of Patients Achieving Response (Based on CDAI Score)
Description: "Response" is defined as the reaction to a stimulus or to a treatment, especially in a favorable way.
  CDAI (Crohn's Disease Activity Index): frequently used to assess disease severity. It gives a score ranging from 0 to over 600, based on a diary of symptoms kept by the patient for 7 days, and other measurements such as the patient's weight and haematocrit.
  The higher the score, the worse is patient's situation. A patient is defined 'remissed' whether the CDAI score is lower than 150 points.
  A patient is defined 'responder' whether the change in CDAI score versus baseline is greater to 100 points
Time Frame: Weeks 4 and 8, and follow-up at 1 month
Population: ITT population included all randomized patients who took at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ITF2357
Number analyzed (Participants) | 26 | 25
Participants
  At week 4 | 11 | 6
  At week 8 | 14 | 8
  At follow up, after one month | 14 | 11

10. Secondary Outcome: Number of Patients With at Least One Related Adverse Event to Study Treatment
Description: Treatment-related adverse events are adverse events (AE) which occurs during an interventional study and which are surely related to study treatment dosing.
Time Frame: At Pre-Treatment period (Week 0); At treatment period (Week 1, Week 2, Week 4, week 6, Week 8); At Follow-up period (1month)
Population: ITT population includes all randomized patients who took at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ITF2357
Number analyzed (Participants) | 26 | 25
Participants | 13 | 12

11. Secondary Outcome: Plasma Levels of ITF2357 Before Morning Dose of ITF2357
Description: Individual plasma levels of ITF2357 (before morning dose) after repeated oral administration of ITF2357 (50mg b.i.d.) in patients with Crohn's disease were assessed.
Time Frame: Pre-dose, week 2, week 4, week 6
Population: Per Protocol Population (PP) - all randomized patients who received at least one dose of study medication without major protocol deviations
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ITF2357
Number analyzed (Participants) | 21
ng/mL
  Pre-dose | 0.00 (0.00)
  Week 2 | 16.87 (6.09)
  Week 4: number analyzed (Participants) | 20
  Week 4 | 16.97 (11.54)
  Week 6: number analyzed (Participants) | 17
  Week 6 | 14.50 (6.78)

12. Secondary Outcome: Plasma Levels of Metabolite ITF2374 Before Morning Dose of ITF2357.
Description: Individual plasma levels of metabolite ITF2374 (before morning dose) after repeated oral administration of ITF2357 (50mg b.i.d.) in patients with Crohn's disease were assessed.
Time Frame: Pre-dose, week 2, week 4, week 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ITF2357
Number analyzed (Participants) | 21
ng/mL
  Pre-dose | 0.00 (0.00)
  Week 2 | 15.09 (6.92)
  Week 4 | 12.93 (7.36)
  Week 6 | 13.24 (8.16)

13. Secondary Outcome: Plasma Levels of Metabolite ITF2375 Before Morning Dose of ITF2357.
Description: Individual plasma levels of Metabolite ITF2375 (before morning dose) after repeated oral administration of ITF2357 (50mg b.i.d.) in patients with Crohn's disease were assessed.
Time Frame: Pre dose, week 2, week 4, week 6.
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ITF2357
Number analyzed (Participants) | 21
ng/mL
  pre-dose | 0.00 (0.00)
  week 2 | 121.23 (88.83)
  week 4 | 112.80 (109.74)
  week 6 | 101.36 (76.32)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Week 0 up to week 8 and during follow up period (which lasts for one month)
Arm/Group | Placebo | ITF2357
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/26 | 3/25
Other Adverse Events (participants affected / at risk) | 17/26 | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | ITF2357 (N=25)
Crohn's Disease (Gastrointestinal disorders) | 1 (1) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | ITF2357 (N=25)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 5 (5)
Crohn's disease (Gastrointestinal disorders) | 3 (3) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Perianal Erythema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal Abscess (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces Discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pruritus Ani (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Chest Pain (General disorders) | 0 (0) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (2)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Rotavirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0)
Blood Magnesium decreased (Investigations) | 1 (1) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
pH Urine increased (Investigations) | 1 (1) | 0 (0)
Red blood cell sedimentation rate increased (Investigations) | 1 (1) | 0 (0)
Sputum Abnormal (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1)
Micturition Disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Bacteriuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Systolic Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No